CLINICAL TRIAL: NCT04247776
Title: Prehabilitation for Colorectal Surgery: A Pragmatic Effectiveness-Implementation Randomized Controlled Trial
Brief Title: Pragmatic Prehabilitation for Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Chelsia Gillis, PhD Candidate, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB18-0979
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Prehabilitation; Colorectal Surgery; Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: Pragmatic RCT Effectiveness- Implementation Hybrid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehab (Experimental): General nutrition, relaxation, and exercise instructions. Home-based functional exercises, Fitbit goals, and nutrition supplements.
  Interventions: Combination Product: Prehab; Other: ERAS; Behavioral: Fitbit
- ERAS (Active Comparator): Enhanced Recovery After Surgery standard of care plus Fitbit.
  Interventions: Other: ERAS; Behavioral: Fitbit

INTERVENTIONS:
Combination Product: Prehab — Exercise: functional exercises, walking, Fitbit goals Nutrition: handout, supplements (protein, vitamins, minerals) Stress reduction: deep breathing
  Arms: Prehab
Other: ERAS — Enhanced Recovery After Surgery guidelines are applied.
Behavioral: Fitbit — Fitbit is worn to monitor step counts.

SUMMARY:
Colorectal surgery is a common surgery for the treatment of colon and rectal cancers as well as other bowel diseases. Recovery from colorectal surgery is difficult because of the many potential negative side effects. These side effects include surgical complications, infections, and long hospital stays. It usually takes several months for patients to recover the strength required to return to their typical daily activities.

The Enhanced Recovery After Surgery program was established in Alberta in 2013 and uses several strategies to improve short-term patient recovery, including earlier discharge from hospital. Whether the ERAS program also improves long-term patient recovery, including quality of life and return to activities of daily living, is unclear. Whether the ERAS program would benefit from the addition of a prehabilitation element is unclear.

Prehabilitation programs are designed to use the waiting period before colorectal surgery to better prepare patients emotionally and physically for their operation. To date, successful prehabilitation programs have used a personalized care strategy where each patient is provided specific care instructions by healthcare professionals to meet their unique exercise, nutrition, and psychological needs. This prehabilitation strategy has been criticized for not being sustainable in our healthcare system.

A new prehabilitation program in response to this criticism is proposed. The prehabilitation program will be conducted in a more sustainable way by offering the program as a group class with a home-based component. ERAS patients at the Peter Lougheed Center are already offered a group class as part of the standard ERAS program. The prehabilitation class will be an extension of this group class that provides general nutrition, exercise, and anxiety-reduction/relaxation strategies to help patients prepare physically and emotionally for their operation. At this class, patients will learn to eat well, practice deep breathing exercises for relaxation, perform simple functional exercises, and to walk for exercise before their surgery. The surgical experience and outcomes of patients who received the additional prehabilitation care will be compared to those who received ERAS care only.

The overall goal of the study is to better understand how ERAS supports recovery after surgery and whether a prehabilitation program offers any additional benefits to the ERAS program currently in place.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* elective colorectal surgery for primary disease under ERAS care at PLC;
* have at least two weeks to participate before their scheduled surgery (i.e., surgery will NOT be rescheduled based on participation in this program);
* are able to walk;
* sufficient fluency in English to complete questionnaires.

Exclusion Criteria:

* emergent surgery;
* dairy allergy;
* galactosemia;
* strict vegans;
* presence of a condition that could compromise the safety of the patient or adherence to the program, including

  * Co-morbid medical, physical, and/or mental conditions including dementia, disabling orthopedic and neuromuscular disease, psychosis;
  * Severe cardiopulmonary abnormalities, sepsis, and end-stage organ disease: cardiac failure (New York Heart Association classes III-IV), chronic obstructive pulmonary disease, renal failure (creatinine > 115µmol/l), hepatic failure (liver aminotranferases >50% the normal range).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Length of stay (LOS) | from date of surgery until hospital discharge, recorded in days, and assessed up to 6 weeks post-surgery
  Length of hospital stay

SECONDARY OUTCOMES:
Complications | from date of surgery until 30 days post-surgery
  Any complication within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chelsia Gillis, PhD(c), Principal Investigator — University of Calgary
Locations (1):
- Peter Lougheed Center, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillis C, Li C, Lee L, Awasthi R, Augustin B, Gamsa A, Liberman AS, Stein B, Charlebois P, Feldman LS, Carli F. Prehabilitation versus rehabilitation: a randomized control trial in patients undergoing colorectal resection for cancer. Anesthesiology. 2014 Nov;121(5):937-47. doi: 10.1097/ALN.0000000000000393. PMID 25076007
- [Background] Gillis C, Fenton TR, Sajobi TT, Minnella EM, Awasthi R, Loiselle SE, Liberman AS, Stein B, Charlebois P, Carli F. Trimodal prehabilitation for colorectal surgery attenuates post-surgical losses in lean body mass: A pooled analysis of randomized controlled trials. Clin Nutr. 2019 Jun;38(3):1053-1060. doi: 10.1016/j.clnu.2018.06.982. Epub 2018 Jul 9. PMID 30025745
- [Background] Gillis C, Buhler K, Bresee L, Carli F, Gramlich L, Culos-Reed N, Sajobi TT, Fenton TR. Effects of Nutritional Prehabilitation, With and Without Exercise, on Outcomes of Patients Who Undergo Colorectal Surgery: A Systematic Review and Meta-analysis. Gastroenterology. 2018 Aug;155(2):391-410.e4. doi: 10.1053/j.gastro.2018.05.012. Epub 2018 May 8. PMID 29750973
- [Derived] Gillis C, Hasil L, Keane C, Brassard D, Kiernan F, Bellafronte NT, Culos-Reed SN, Gramlich L, Ljungqvist O, Fenton TR. A multimodal prehabilitation class for Enhanced Recovery After Surgery: a pragmatic randomised type 1 hybrid effectiveness-implementation trial. Br J Anaesth. 2025 Apr 7:S0007-0912(25)00153-9. doi: 10.1016/j.bja.2025.03.001. Online ahead of print. PMID 40199628